| Official Title: | A Single-Arm, Open-Label, Phase I/II Study of Glasdegib |
|-----------------|---------------------------------------------------------|
| | for Sclerotic Chronic Graft-vs-Host Disease |
| NCT Number: | NCT04111497 |
| Document Type: | Informed Consent Form |
| Date of the | 6/9/2022 |
| Document: | |

#### Fred Hutchinson Cancer Research Center

## Consent to take part in a research study:

# A Single-Arm, Open-Label, Phase I/II Study of Glasdegib for Sclerotic Chronic Graft-vs-Host Disease

Principal Investigator: Stephanie Lee, MD, MPH. University of Washington; Fred Hutchinson Cancer Research Center. 206-667-5160

## Emergency number (24 hours): (206) 598-8902

Ask to page the Long-Term Follow-Up Attending

### Important things to know about this study.

You are invited to participate in a research study. The purpose of this research is to see if a medication called glasdegib (Daurismo<sup>TM</sup>) is helpful in treating skin thickening that can happen as part of chronic graft-versus-host disease (GVHD).

People who agree to join the study will be asked to attend up to 18 visits over 24 months. The study involves taking an oral medication (glasdegib) and attending regular study visits for physical exams, blood draws, lung function testing, and other assessments.

We do not know if glasdegib will help treat chronic GVHD, and it could even make your condition/disease worse. Glasdegib could cause side effects such as low blood counts, muscle spasms, and kidney impairment, as described below in this form.

You do not have to join this study. You can choose to receive standard methods to treat chronic GVHD instead of participating in this study. We will give you details about the purposes, procedures, risks and possible benefits related to this study. We will explain other choices that you have. We will also give you any other information that you need in order to make an informed decision about joining this study.

The following is a more complete description of this study. Please read this description carefully. You can ask any questions you want to help you decide whether to join the study. If you join this study, we will give you a signed copy of this form to keep for future reference.

## We invite you to join this research study.

We invite you to join this research study because you have skin thickening and/or joint tightening caused by chronic GVHD, and it has not responded to at least one prior medication. Up to 20 people will join this study.

Research is not the same as treatment or medical care. The purpose of a research study is to answer scientific questions.

You do not have to be in the study. You are free to say "yes" or "no", or to drop out after joining. If you say "no," you would have no penalty or loss of benefits. Whatever you decide, your regular medical care would not change.

## Why are we doing this study?

We are doing this study to see if glasdegib is helpful in the treatment of chronic GVHD. The study will enroll people who have active GVHD-related sclerosis or fasciitis despite at least one prior chronic GVHD treatment.

In this study, we want to learn what effects, good or bad, glasdegib has on people with chronic GVHD. If you join this study, we would give you glasdegib and watch carefully for any side effects.

## What research tests, procedures, and treatments are done in this study?

If you join this study, we would do these tests and procedures:

- Questionnaire We would ask you to fill out five questionnaires—one
  when you start taking glasdegib, then one every three months, plus
  one more when you finish treatment. Each questionnaire has questions
  about your GVHD symptoms and general health. Some of the
  questions may be sensitive. You can choose not to answer any
  questions that make you feel uncomfortable.
- Physical exam You will have a physical exam at each study visit, and we will pay special attention to any signs or symptoms of GVHD that you may be having. A member of the study team will fill out a form about your GVHD.
- Clinical labs We will do blood tests to check for GVHD and overall health. Most of the time, these labs will be done as part of your normal medical care.
- Research blood samples We will collect 24 ml (about 1.5 tablespoons) of blood four times for research.
- **Electrocardiogram** We will perform an electrocardiogram (ECG) fourteen times during the study to check your heart rate and rhythm.
- Pulmonary function test and spirometry When you enroll on the study, we will do full pulmonary function tests, which checks how well

your lungs work. Eight more times during the study, we will ask you to do just the spirometry part of the test, which involves blowing into a small hand-held device.

- Skin biopsies Before you start taking glasdegib, and about 6
  months later, we will ask if we can take a skin biopsy for research. This
  is optional and you can still be in the study if you decide not to do the
  biopsies.
- Pregnancy test If you are a woman of childbearing potential, we will
  do a blood test to check for pregnancy before you begin taking
  glasdegib.

If you need to stop taking glasdegib early, we would still ask you to complete the study visits and assessments at 3, 6, 9, 12, 15, 18, 21 and 24 months unless you start a new medication for chronic GVHD. After about two years of active study participation, you would no longer have study visits, but we would still like to follow your health and GVHD by looking at your medical records periodically.

## How long would you stay in this study?

If you join this study, you would have study visits for about 26 months. After that, we would continue to look at your medical records periodically.

You would receive glasdegib for up to 24 months. After your last dose of glasdegib, you would have a follow-up exam about one month later.

Doctors could take you out of this study at any time. This would happen if:

- They think it is in your best interest not to continue in the study.
- You are not able or willing to follow study procedures.
- You start a new medication for your chronic GVHD.
- The whole study is stopped.

If you withdraw from the study for any reason, previously collected information would remain in the study records and would be included in the analysis of results. This information could not be removed from the study records.

**Long-term follow-up** means keeping track of someone's medical condition for a long time. If you join this study, we would review your medical records a few times per year to see how you are doing. If you are not seen at the study center, we might also ask your local doctor to send a copy of your medical records. This information will help us learn about the long-term effects of glasdegib and chronic GVHD treatment in general.

You do not have to be in long-term follow-up. You could say "yes" or "no". Either way, you could still join this study. If you drop out of the study, you would be asked if we could continue to review your medical records.

If you choose not to join long-term follow-up, you would not be contacted regularly, and we would not ask your doctor to send medical records, but we might still need to contact you for some other reason.

## What are the side effects (risks)?

In this part of the consent form, we describe the side effects we expect from the tests and treatments in this study. Glasdegib could cause side effects we do not know about yet. We will carefully watch everyone in the study for side effects.

If you join this study, we would tell you if we discover new side effects that could affect you.

This form lists the most common side effects of glasdegib. Other side effects could occur when glasdegib is used together with other drugs.

Side effects may be mild or very serious. Medicines could be given to help lessen side effects. Many side effects go away soon after you stop taking glasdegib. In some cases, side effects can last a long time or never go away. There also is a risk of death with any medication.

## Low cell counts (cytopenias)

Low cell counts can make you get infections more easily and can cause low energy. We will monitor your blood counts during the study to watch for this complication.

## **Heart rhythm changes (QT/QTc prolongation)**

This can be seen in people who already have heart disease, or who are taking other medications that also affect their heart rhythm. We will do electrocardiograms to watch for this complication.

#### **Kidney impairment**

Some people who take glasdegib have decreased kidney function, and this usually happens in patients who already have a risk of kidney problems. We will monitor your kidney function with blood tests during the study.

#### Muscle spasms or cramps

Some people who take glasdegib experience muscle spasms or cramps. These cramps might be severe enough to interfere with your daily activities or sleep. If this happens, please tell your study doctor right away.

#### Low sodium (hyponatremia)

We will monitor your blood levels of sodium during the study.

## Taste changes (dysgeusia)

This is a common side effect with glasdegib and is usually not bad enough to make people stop taking glasdegib. If you have taste changes that are bothersome, please tell the study doctor.

## Hair loss (alopecia)

Some people notice hair loss when they are taking glasdegib. Please tell your study doctor if you notice new hair loss.

#### **Dental effects**

Glasdegib has been associated with loose teeth and toothache in some studies. You should see your dentist regularly and report any symptoms.

## Reproductive risks

Taking glasdegib involves risks to an embryo, fetus (unborn baby) or nursing infant; it can cause the child to die before it is born (be stillborn) or have severe birth defects. Therefore, you could not join this study if you are pregnant, if you are planning to become pregnant, or if you are breast-feeding.

If you became pregnant after joining this study, you would have to notify the study doctor immediately. Participation in this study would end, and you would receive counseling and follow-up throughout the pregnancy and for about 6 months after the child is born.

#### For females who can become pregnant:

- You should talk to the study doctor about the risks of glasdegib to your unborn child.
- You will be asked to undergo a pregnancy test within 7 days before you start glasdegib.
- You should not use glasdegib during pregnancy.
- You should use effective birth control during treatment and for at least 30 days after your last dose of glasdegib. Talk with the study doctor about what birth control method is right for you during this time. If you are already using a method of birth control, you would have to check with the study doctor or a member of the study staff to make sure it is acceptable.
- Talk to the study doctor right away if you have unprotected sex or if you think that your birth control has failed.
- Tell the study doctor right away if you become pregnant or think that you may be pregnant.

#### For males:

- It is not known if glasdegib is present in semen. Do not donate semen during treatment with glasdegib and for at least 30 days after your last dose.
- You should always use effective birth control, including a condom, even if you have had a vasectomy, during sex with female partners who are pregnant or who are able to become pregnant, during treatment with glasdegib and for at least 30 days after your last dose to protect your female partner from being exposed to glasdegib.
- Tell the study doctor right away if your partner becomes pregnant or thinks she is pregnant while you are taking glasdegib.

## **Exposure to glasdegib during pregnancy:**

If you think that you or your female partner may have been exposed to glasdegib during pregnancy, tell the study doctor right away. If you become pregnant during treatment with glasdegib, you or the study doctor would need to report your pregnancy to Pfizer at 1-800-438-1985.

## Other risks involved with the study

- The blood draw may briefly cause you to feel faint, lightheaded, or nauseated. There is a risk of bleeding, bruising, and rarely, infection.
- There is a risk of discomfort, bleeding, infection, and scarring from the optional skin biopsies.
- The breathing tests can cause you to cough or feel lightheaded.
- The survey questions we ask about your symptoms and quality of life may make you feel uncomfortable. You can skip any question you do not want to answer.
- There is a slight risk of loss of confidentiality.

#### What are the benefits?

We do not know if this study would help you. We are testing glasdegib to see its effects on people with chronic GVHD, and to find the safest dose in people with chronic GVHD. You might get better if you receive glasdegib, but your condition could stay the same or even get worse. We hope the information from this study will help other people with chronic GVHD in the future.

## You have other choices besides this study.

You do not have to join this study. You are free to say "yes" or "no". Your regular medical care would not change if you decide to say "no".

You have other choices for treatment. Each of these choices has risks and benefits. You should talk to your doctor or healthcare provider about these choices.

Your other choices may include:

- Continue routine treatment or care for your cGVHD without being in a clinical study
- Ibrutinib, an FDA approved drug for the treatment of cGVHD if you have had at least one prior line of therapy
- Take part in another clinical study
- No treatment

Enrollment in this study may exclude you from other research studies.

## Protecting Privacy as an Individual and the Confidentiality of Personal Information

If you join this study, some people or organizations might need to look at your medical records and research records for quality assurance or data analysis. They include:

- Researchers involved with this study.
- Pfizer and their agents.
- Institutional Review Boards (IRB), including the Fred Hutchinson Cancer Research Center IRB. An IRB is a group that reviews the study to protect the rights and welfare of research participants.
- Fred Hutchinson Cancer Research Center, University of Washington, and Seattle Cancer Care Alliance.
- Office for Human Research Protections, Food and Drug Administration, and other regulatory agencies as required.

We will do our best to keep personal information confidential. But we cannot guarantee total confidentiality. Personal information may be given out if required by law. For example, workplace safety rules may require health workers to contact you about lab tests. Or a court may order study information to be disclosed. Such cases are rare.

We will not use personal information in any reports about this study, such as journal articles or presentations at scientific meetings.

If you join this study, information about your participation would be made part of your permanent medical record. This information would include a copy of this consent form. If an insurance company or employer or anyone else were

authorized to see your medical record, they would see a copy of this consent form.

## How is my genetic information protected?

A federal law called the Genetic Information Nondiscrimination Act (GINA) helps protect genetic information about people who join research studies.

GINA restricts access to genetic information so that it cannot be used for health insurance coverage decisions. GINA prevents health insurance companies or group health plans from:

- Asking for genetic information obtained in research studies, or
- Using genetic information when making decisions regarding your eligibility or premiums

GINA *does not* help or protect against genetic discrimination by companies that sell life, disability or long-term care insurance.

## Would we pay you if you join this study?

There is no payment for being in this study.

## Would you have extra costs if you join this study?

You or your insurance company will not be billed for tests and procedures done specifically for this study (i.e., extra blood drawn for research, pregnancy tests, or questionnaires). Glasdegib will be provided free of charge from Pfizer for up to 24 months.

There are some extra costs for being in this study. You or your insurer will have to pay these costs. Some insurers will not pay for research. Check with your insurer before you join this study.

#### The extra costs are:

- Cost of tests that are given more often than usual.
- Cost of standard doctor visits and lab tests.
- Cost of any other medical care you may need because of this study.

Whether you are in the study or not, you or your insurance company will be responsible for medications, tests, clinic and hospital visits as part of your routine care as a transplant recipient. Pfizer will not pay any money to you or pay any of your medical bills.

## What if you get sick or hurt after you join this study?

For a life threatening problem, call 911 right away or seek help immediately. Contact your study doctor when the medical emergency is over or as soon as you can.

For all other medical problems or illness related to this research, immediately contact Dr. Lee at 206-667-5160. She will treat you or refer you for treatment. You or your health insurance will have to pay for the treatment. There are no funds to pay you for a research-related injury, added medical costs, loss of a job, or other costs to you or your family. State or national law may give you rights to seek payment for some of these expenses. You do not waive any right to seek payment by signing this consent form.

You or your insurer will be billed for treatment of problems or complications that result from your condition or from standard clinical care.

You would not lose any legal right to seek payment for treatment if you sign this form.

## What will my information and/or tissue samples be used for?

Your information and tissue samples (such as blood and skin biopsies) will be used for the purposes of this study.

Your tissue samples might help researchers develop new products. This research could be done by for-profit companies. There is no plan to share with you any revenue generated from products developed using your tissue samples.

During this study, if the researchers learn new information that may be important to your general health or to your disease or condition, they will share that information with you. For example, if your physical exam, clinical blood tests, ECG, or pulmonary function tests show abnormalities, we would discuss those with you. The research blood samples and optional skin biopsies will be stored and analyzed later. The results of any testing on those samples would not be available to you.

In addition, be aware that by agreeing to participate in this study, your information or tissue samples could be used for future research studies or sent to other investigators for future research studies without additional consent from you. These future research studies will be reviewed by an oversight group known as an institutional review board if required by law. The information that identifies you will first be removed from your information or tissue samples. If you do not want your information or tissue samples to be used for future research studies without your consent, you should not participate in this study.

#### We invite you to donate tissue samples for other research.

After we do tests on tissue (blood or skin) in this study, some tissue may be left over. We invite you to donate this leftover tissue for future research. This may include genetic research.

If you join this study, you would not have to donate tissue for future research. You would be free to say "yes" or "no." Regular medical care would not change if you say "no."

If you donate tissue, it would be stored in a secure location. If we want to use your tissue for other research or share it with other scientists for research, an ethics review committee (IRB) would review the request. The IRB would decide if we need to ask you for permission to do the research.

Your donated tissue would be used only for research. This research could be done by for-profit companies. Researchers would not report their results to you or your doctors. The research results would not be included in medical records. The results would not affect your medical care.

Research with tissue might help develop new products. If these products make money, there is no plan to share the money with the participants who donate the tissue.

If you donate tissue for research, you could withdraw the donation at any time by calling Dr. Stephanie Lee at 206-667-5160. You would have no penalty for withdrawing the donation, and regular medical care would not change. We could not return donated tissue, but we might be able to destroy the donated tissue. We could not destroy tissue if it is stored or shared without any label saying who donated it. In this case, it could still be used for research.

## Your rights

- You do not have to join this study. You are free to say "yes" or "no".
- If you get sick or hurt in this study, you do not lose any of your legal rights to seek payment by signing this form.
- During the study, we might learn new information that you need to know. For example, some information may affect your health or wellbeing. Other information might make you change your mind about being in this study. If we learn these kinds of information, we would tell you.
- If you join this study, you would not have to stay in it. You could stop at any time (even before you start). Your regular medical care would not change. You would have no penalty for stopping, but it would be better not to join the study if you think that you would change your mind later.

- If you decide to drop out, we would want you to tell the study doctor.
  The doctor could tell you about the effects of stopping glasdegib. You
  and the doctor could talk about the follow-up care and testing that
  would help the most.
- Before you leave the study, the doctor might ask you to continue in the follow-up part of the study (we would review your medical records periodically).

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

## Your responsibilities

If you join this study, you would have some responsibilities.

- Follow the schedule of study visits and procedures.
- Take study medications as directed.
- Prevent pregnancy.
- Tell us about side effects.

#### For more information

If you have questions or concerns about this study, you can talk to your doctor anytime. Other people you could talk to are listed below.

| If you have questions about: | Call: |
|---|---|
| This study (including complaints and requests for information) | (206) 667-6190 (Dr. Stephanie Lee)<br>(206) 667-7010 (Research Coordinator) |
| If you get sick or hurt in this study | (206) 667-6190 (Dr. Lee) |
| Your rights as a research participant | 206-667-5900 or email irodirector@fredhutch.org (Director of Institutional Review Office, Fred Hutchinson Cancer Research Center) |
| Your bills and health insurance coverage | (206) 606-6226 or toll free at (800) 804-8824 |

## Emergency number (24 hours): (206) 598-8902

Read each question and think about your choice. When you decide on each question, please circle **YES** or **NO**.

Do you agree to donate your leftover tissue for future studies of GVHD?

(circle one)

YES

NO

## **Signatures**

Please sign below if you:

- have read this form (or had it read to you);
- had the opportunity to ask any questions you have;
- had the opportunity to discuss the research with the person obtaining consent; and
- agree to participate in this study.

Previous consent version date: 17-Dec-2019 Copies to: research coordinator, HIM, patient

| Participant: | | |
|---|---|---|
| Printed Name | Signature | Date |
| Researcher's statement | | |
| | esearch study, including proce<br>A copy of the signed consent | |
| Person obtaining conser | nt signature: | |
| Printed Name | Signature | Date |
| Protocol: 8771<br>Current consent version da | nte: 09-Jul-2020 | |